CLINICAL TRIAL: NCT00935922
Title: CCRC: Understanding the Effects of Omega-3 Fatty Acids vs. Lignans in Flaxseed on Metabolic and Inflammatory Markers Leading to Diabetes and Cardiovascular Disease.
Brief Title: CCRC: Understanding the Effects of Omega-3 Fatty Acids Versus Lignans in Flaxseed on Metabolic and Inflammatory Markers Leading to Diabetes and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Flax Canada 2015 Inc. (Industry)
Responsible Party: Principal Investigator, Sidika E. Karakas, MD, Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 200816799-1
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2009-07

CONDITIONS: Body Weight; Lipids; Blood Glucose; Insulin
Keywords: Flaxseed; Weight loss; Heart health; Diabetes
MeSH Terms: conditions — Body Weight; Insulin Resistance; Weight Loss; Diabetes Mellitus | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Soybean oil bar (Placebo Comparator): A nutrition bar enriched with soybean oil
  Interventions: Dietary Supplement: Flaxseed
- Flaxseed bar with low lignans (Experimental): A nutrition bar enriched with flaxseed oil
  Interventions: Dietary Supplement: Flaxseed
- Flaxseed bars with high lignans (Experimental): A nutrition bar enriched with flaxseed oil and high lignans
  Interventions: Dietary Supplement: Flaxseed

INTERVENTIONS:
Dietary Supplement: Flaxseed — Flaxseed omega-3 fatty acids and lignans

SUMMARY:
The aim of this study is to compare the effects of flaxseed on atherogenic lipids, plasma inflammatory markers, and insulin sensitivity.

We hypothesize that flaxseed omega-3 fatty acids will improve the lipid profile (decrease triglyceride, total and LDL-cholesterol and increase HDL-cholesterol).

Flaxseed is the richest dietary source of lignan secoisolariciresinol diglucoside (SDG). Lignans are estrogens found in plant sources that behave similar to endogenous estrogens and have been associated with cardiovascular benefits due to their antioxidant activity. Therefore, we also hypothesize that flax-lignans will cause a significant decrease in LDL oxidation and in inflammatory markers such as C-reactive protein (CRP), interleukin-6 (IL-6), IL-1B, serum fatty acid binding protein 4 (FABP-4), and serum amyloid attached to high density lipoprotein (HDL-SAA).

ELIGIBILITY:
Inclusion Criteria:

* Men or postmenopausal women in the 40-65 years age range. Body Mass Index in the range of 25-39

Exclusion Criteria:

* Women are are premenopausal
* Smoking
* Diabetes
* Cancer
* Gout
* Untreated thyroid disease
* Kidney Disease
* Liver Disease
* Use of lipid lowering drugs
* Use of insulin sensitizing drugs
* Use of ACE inhibitors or other blood pressure lowering medications
* Use of over the counter or prescription anti-obesity medications
* Weight loss of 10% or more within the last 12 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Improved lipid profile | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sidika Kasim-Karakas, MD, Principal Investigator — University of California, Davis Health System
Locations (1):
- CCRC, Mather, California, United States